CLINICAL TRIAL: NCT01911429
Title: A 6-Week Randomized, Parallel, Double-Blind, Placebo-Controlled, Fixed-Dose, Multicenter Study To Evaluate The Efficacy and Safety of Lurasidone in Adolescent Subjects With Schizophrenia
Brief Title: Pediatric Schizophrenia Efficacy and Safety Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1050301; 2013-001695-38 (EudraCT Number)
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Lurasidone; Latuda
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lurasidone 40 mg (Experimental): Lurasidone 40 mg once daily
  Interventions: Drug: Lurasidone 40 mg
- Lurasidone 80 mg (Experimental): Lurasidone 80 mg once daily Arm received the Lurasidone 40mg dose first, from Days 1-3, and then received the Lurasidone 80 mg dose from day 4 to Week 6
  Interventions: Drug: Lurasidone 80 mg
- Placebo (Placebo Comparator): Placebo 40 or 80 mg once daily
  Interventions: Drug: Placebo 40 or 80 mg

INTERVENTIONS:
Drug: Lurasidone 40 mg — Lurasidone 40 mg once daily
  Other Names: Latuda
  Arms: Lurasidone 40 mg
Drug: Lurasidone 80 mg — Lurasidone 80 mg once daily
  Other Names: Latuda
  Arms: Lurasidone 80 mg
Drug: Placebo 40 or 80 mg — Placebo 40 or 80 mg once daily
  Arms: Placebo

SUMMARY:
Efficacy and Safety study of Lurasidone in pediatric patients.

DETAILED DESCRIPTION:
To evaluate the efficacy of lurasidone (40 mg/day and 80 mg/day) compared with placebo in adolescent subjects with schizophrenia (diagnosed by Diagnostic and Statistical Manual of Mental Disorders, 4th Ed., Text Revision [DSM-IV-TR] criteria) as measured by the change from Baseline in the Positive and Negative Syndrome Scale (PANSS) total score at Week 6.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent(s) or legal guardian(s) with sufficient intellectual capacity to understand the study and support subjects' adherence to the study procedures must be obtained for subjects who are not emancipated. In accordance with Institutional Review Board (IRB) requirements, the subject will complete an informed assent prior to study participation.
* Male or female subjects 13 to 17 years of age, inclusive, at the time of consent.
* DSM-IV-TR axis I primary diagnosis of schizophrenia (including disorganized (295.10), paranoid (295.30), undifferentiated (295.90) subtypes) and confirmation of the schizophrenia diagnosis by an adequately trained clinician at the time of screening, by means of the Schedule for Affective Disorders and Schizophrenia for School-age Children (K-SADS-PL).
* PANSS total score ≥ 70 at screening and Baseline.
* CGI-S ≥ 4 at screening and Baseline.
* Within 5th to 95th percentile for gender specific weight-for-age and height-for-age Growth Charts from National Center for Health Statistics.
* In good physical health on the basis of medical history, physical examination, and laboratory screening.
* Females who participate in this study:

are unable to become pregnant (eg, premenarchal, surgically sterile, etc.); -OR-

practices true abstinence (consistent with lifestyle) and must agree to remain abstinent from signing informed consent to at least 30 days after the last dose of study drug has been taken;

-OR-

are sexually active and willing to use a medically effective method of birth control (e.g., male using condom and female using condom, diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from signing informed consent to at least 7 days after the last dose of study drug has been taken.

* Males must be willing to remain sexually abstinent (consistent with lifestyle) or use an effective method of birth control (eg, male using condom and female using condom, diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from signing informed consent to at least 30 days after the last dose of study drug has been taken.
* In the judgement of the clinician, the subject has an acute exacerbation of psychotic symptoms (no longer than 2 months in duration) and marked deterioration of function from baseline (by history) or, the subject has been hospitalized for the purpose of treating an acute psychotic exacerbation for 2 consecutive weeks or less immediately before screening.
* In the judgment of the investigator, the subject is able to swallow the size and number of study drug tablets specified per protocol.
* Willing and able to adhere to protocol-specified meal requirements during dosing.

Exclusion Criteria:

* Has an Axis I or Axis II diagnosis other than schizophrenia that has been the primary focus of treatment within 3 months of screening.
* Has a history or current diagnosis of mental retardation, neuroleptic malignant syndrome, or any neurologic disorder, or severe head trauma.
* Lifetime history of human immunodeficiency virus (HIV) positive or acquired immune deficiency syndrome (AIDS), or history of Hepatitis B or C.
* Any of the following:

Documented history of chromosomal disorder with developmental impairment (ie, trisomy chromosome 21; 22q11 deletion syndrome).

Evidence of any chronic organic disease of the CNS such as tumors, inflammation, active seizure disorder, vascular disorder, potential CNS related disorders that might occur in childhood- eg, Duchenne Muscular dystrophy, myasthenia gravis, or other neurologic or serious neuromuscular disorders. In addition, subjects must not have a history of persistent neurological symptoms attributable to serious head injury. Past history of febrile seizure, drug-induced seizure, or alcohol withdrawal seizure is not exclusionary.

* PANSS total scores ≥ 120 at screening or Baseline.
* Exhibits evidence of moderate or severe extrapyramidal symptoms, dystonia, tardive dyskinesia, or any other moderate or severe movement disorder. Severity to be determined by the investigator.
* Lifetime history of electroconvulsive therapy (ECT).
* Resistant to antipsychotic treatment based on at least two different prior adequate trials (ie, adequate dose and duration) of an antipsychotic agent within the current episode of schizophrenia.
* Clinically significant neurological, metabolic (including type 1 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, carcinoma, and/or urological disorder that would pose a risk to the subjects if they were to participate in the study or that might confound the results of the study.

Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted. Any subject with a known cardiovascular disease or condition (even if controlled) must be discussed with the Medical Monitor during screening.

* Has a history of malignancy < 5 years prior to signing the informed consent.
* Clinically significant finding(s) on physical examination determined by the investigator to pose a health concern to the subject while on study.
* Clinically relevant abnormal laboratory values or abnormal vital sign values/findings.

Note: If any laboratory results are outside the normal range, the site may have the subject retested. If upon retesting the value remains outside the normal range, the significance of this value must be discussed with the Medical Monitor for enrollment consideration.

* A history or presence of abnormal ECG, which in the investigator's opinion is clinically significant. Abnormal screening ECGs will be centrally over-read, and eligibility will be determined based on the over-read.
* Presence or history (within the last year) of a medical or surgical condition (eg, gastrointestinal disease) that might interfere with the absorption, metabolism, or excretion of orally administered lurasidone.
* Clinically significant alcohol abuse/dependence or drug abuse/dependence based on DSM-IV-TR criteria within the last 6 months prior to screening.
* Positive test results at screening or Baseline for:

  1. Urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine, cannabinoids, and methadone). A positive test for amphetamines, barbiturates, opiates, benzodiazepines or methadone may not result in exclusion of subjects if the investigator determines that the positive test is as a result of taking prescription medicine(s) as prescribed. In the event a subject tests positive for cannabinoids (tetrahydrocannabinol) or alcohol, the investigator will evaluate the subject's ability to abstain from prohibited substances during the study. If in the investigator's clinical judgment the subject will abstain, the subject may be enrolled after consultation with the Medical Monitor.
  2. Pregnancy test.
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* Participated in another interventional clinical trial or receiving an investigational product within 30 days prior to randomization.
* Donation of whole blood within 60 days prior to randomization.
* Known history or presence of clinically significant intolerance to any antipsychotic medications including but not limited to angioedema, serotonin or neuroleptic malignant syndromes.
* Clinically relevant history of drug hypersensitivity to lurasidone or any components in the formulation.
* Use of concomitant medications that consistently prolong the QT/QTc interval within 28 days prior to randomization.
* Received depot neuroleptics unless the last injection was at least 1 month or 1 treatment cycle prior to screening, whichever is longer.
* Received treatment with antidepressants, stimulants, or atomoxetine within 3 days prior to randomization, fluoxetine hydrochloride within 21 days of randomization, monoamine oxidase (MAO) inhibitor within 28 days of randomization, or clozapine within 120 days of randomization.
* Use of any antipsychotic medication (other than study drug), carbamazepine, oxcarbazepine, eslicarbazepine acetate, or fluvoxamine, within 3 days prior to randomization (7 days prior to randomization for aripiprazole) and until follow-up.
* Has a prolactin concentration ≥ 100 ng/mL at screening, or has a history of pituitary adenoma.
* At screening or Baseline the subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C-SSRS.
* Subject is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property during the study. Subject has a history of one or more serious suicide attempts (based on the investigator's judgment) in the 3 months prior to screening. Subjects determined to be at risk of suicide or injury, as assessed by the investigator at screening, will be referred for further psychiatric evaluation.
* Adhering to a special diet for the 28 days prior to drug administration (eg, liquid, protein, raw food diet).
* Subject is planning to move during the study, is chronically homeless, or is unable to attend all planned study visits. The Medical Monitor will be consulted for individual cases, as needed.
* Demonstrates a decrease (improvement) of > 25% in the PANSS score between screening and Baseline visits.
* Subject with newly diagnosed Type 2 diabetes during screening. A subject with Type 2 diabetes is eligible for study inclusion if considered clinically stable, which is defined as:

Random (non-fasting) screening glucose is < 200 mg/dl (11.1 mmol/L); and If ≥ 200 mg/dL (11.1 mmol/L) must be retested in a fasted state. Retested fasted value cannot be ≥ 126 mg/dL.

HbA1c ≤ 6.5%; and If a subject is currently being treated with oral anti-diabetic medication(s), the dose must have been stable for at least 4 weeks prior to screening. Such medication may be adjusted or discontinued during the study, as clinically indicated.

* Subject has required hospitalization for diabetes or related complications in the past 12 months.
* Subject requires use of concomitant medications that are potent inducers or inhibitors of the cytochrome P450 (CYP) 3A4 enzyme system (Appendix C) from signing informed consent until follow-up.
* Clinically significant orthostatic hypotension (ie., a drop in systolic blood pressure of 20 mmHg or more and/or drop in diastolic blood pressure of 10 mmHg or more within 4 minutes of standing up).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 327 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lurasidone Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (90):
- United States (36):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - California Pharmaceutical Research Institute, Inc, Anaheim, California
  - Central Valley Medical Research, Bakersfield, California
  - ProScience Research Group, Culver City, California
  - Diligent Clinical Trials, Inc, Downey, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Global Clinical Trials, LLC, Irvine, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Asclepes Research, Panorama City, California
  - CITrials, Inc. - Riverside & San Bernardino County, Riverside, California
  - Hartford Hospital, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials - Parent, Gainesville, Florida
  - APG Research, LLC, Orlando, Florida
  - Medical Research Group of Central Florida, Sanford, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Institute for Behavioral Medicine, LLC, Smyrna, Georgia
  - Baber Research Group, Naperville, Illinois
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Neurobehavioral Medicine Group, PLLC, Bloomfield Hills, Michigan
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Manhattan Behavioral Medicine, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - BioBehavioral Research of Austin, Austin, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - BioBehavioral Research of Austin, El Campo, Texas
  - Family Psychiatry of The Woodlands, P.A., The Woodlands, Texas
  - Aspen Clinical Research, Orem, Utah
  - University of Virginia, Charlottesville, Virginia
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Bulgaria (4):
  - MHC - Ruse, EOOD, Rousse
  - UMHAT "Alexandrovska" EAD, Sofia
  - MHAT-Targovishte, AD, Targovishte
  - MHAT 'Sv. Marina', EAD, Varna
- Colombia (3):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Barranquilla
  - E.S.E. Hospital Mental de Antioquia, Bello
  - Centro de Investigaciones del Sistema Nervioso Limitada - Grupo CISNE Ltda, Bogotá
- France (2):
  - CHU Nantes - Hôpital Mère-Enfant, Nantes, Loire Atlantique
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice
- Hungary (2):
  - Vadaskert Alapitvany a Gyermekek Lelki Egeszsegeert, Budapest
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
- University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur, Malaysia
- Mexico (3):
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Accelerium S. de R.L. de C.V., Monterrey
  - Instituto de Informacion de Investigacion en Salud Mental, Monterrey
- Philippines (4):
  - Alexian Brothers Health and Wellness Center, Daveo City
  - West Visayas State University Medical Center, Iloilo City
  - National Center for Mental Health, Mandaluyong
  - Veterans Memorial Medical Center, Quezon City
- Poland (3):
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - NZOZ Poradnia Zdrowia Psychicznego, Tyniec Mały
  - Instytut Psychiatrii i Neurologii, Warsaw
- Puerto Rico (3):
  - Centro de Investigacion Clinica Psiquiatrica, Caguas
  - Centro de Investigacion Clinica Psiquiatrica, Ponce
  - INSPIRA Clinical Research, San Juan
- Romania (3):
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul Clinic de Psihiatrie Socola, Iași
  - Spitalul Clinic de Urgenta pentru Copii "Louis Turcanu" Timisoara, Timișoara
- Russia (7):
  - Regional Government Institution Kipetsk Regional Psychoneurology Hospital, Lipetsk
  - St. Petersburg State Healthcare Institution (SPSHI), Saint Petersburg
  - FSBI "Bekhterev Psychoneurological Research Institute SPb Russia", Saint Petersburg
  - SHI Regional Clinical Psychiatry Hospital of St. Sofia, Saratov
  - FSBSI "Scientific Research Institute of Mental Health", Tomsk
  - Nizhny Novgorod Regional State Institution of Healthcare, Veliky Novgorod
  - Sverdlov regional Psychiatric Clinical Hospital, Yekaterinburg
- South Korea (3):
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (2):
  - Hospital Marítimo de Torremolinos, Torremolinos, Málaga
  - Hospital Sant Joan de Deu, Barcelona
- Ukraine (10):
  - RPsH #3 Сhildren Dept SHEI Ivano-Frankivsk SMU, Ivano-Frankivsk
  - SI Institute of Neurology, Psychiatry and Narcology of NAMSU, Kharkiv
  - SI Institute of Children and Adolescents Healthcare of NAMSU, Kharkiv
  - CI Kherson Regional Psychiatric Hospital of Kherson RC, Kherson,Vil. Stepanivka
  - TMA Psychiatry in Kyiv Center of NT & Rehabilitation of Psychotic Conditions, Kyiv
  - CI Lviv Regional Clinical Psychiatric Hospital, Lviv
  - CI Odesa Regional Medical Center of Mental Health, Odesa
  - O.F. Maltcev Poltava RCPsH Children Dept Ukrainian Medical Stomatological Academy, Poltava
  - Ternopil RCCPH Dept of Psychiatry #9 (adolescent)& #8 (pediatric) Ternopil I.Ya. Gorbachevskyi SMU, Ternopil
  - M.I. Pyrogov VNMU Ch of Psych&Nar BO CI O.I. Yuschenko VRPsH, Vinnytsia
- United Kingdom (3):
  - Royal Cornhill Hospital, Aberdeen, Strathclyde
  - Northcroft, Birmingham
  - Royal Edinburgh Hospital, Edinburgh

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 80 mg: Lurasidone 80 mg once daily
  Lurasidone 80 mg: Lurasidone 80 mg once daily Subjects received lurasidone 40/mg day from Days 1-3, and 80mg/day from days 4 to Week 6 visit
Period: Overall Study
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Started | 108 | 106 (Subjects received lurasidone 40/mg day from Days 1-3, and 80mg/day from days 4 to Week 6 visit) | 113 (one subject randomized to Placebo group was never dosed for study medication, making the total 112)
Completed | 96 | 96 | 93
Not Completed | 12 | 10 | 20
Not completed — Adverse Event | 5 | 3 | 9
Not completed — Lack of Efficacy | 1 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 5 | 4
Not completed — Accidental randomization | 0 | 0 | 1
Not completed — subject left study | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: two subjects from the lurasidone 80mg (originally 106) group transferred to the lurasidone 40 mg (originally 108) group
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo | Total
Number analyzed (Participants) | 110 | 104 | 112 | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 110 | 104 | 112 | 326
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.33) | 15.3 (1.35) | 15.3 (1.37) | 15.4 (1.35)
Age, Customized [Count of Participants; unit: Participants]
  13-15 years old | 50 | 55 | 55 | 160
  16-17 years old | 60 | 49 | 57 | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 70 | 71 | 208
  Male | 43 | 34 | 41 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 18 | 13 | 44
  Not Hispanic or Latino | 97 | 86 | 99 | 282
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 4 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 18 | 22 | 60
  White | 73 | 73 | 74 | 220
  More than one race | 11 | 9 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 38 | 35 | 37 | 110
  South America | 9 | 8 | 9 | 26
  Europe | 5 | 57 | 61 | 123
  Southeast Asia | 2 | 1 | 1 | 4
  East Asia | 2 | 1 | 1 | 4
Baseline BMI Percentile [Number; unit: participants]
  < 3th percentile | 0 | 1 | 1 | 2
  > 3th to 85th percentile | 74 | 65 | 72 | 211
  >97th percentile | 6 | 6 | 8 | 20
Baseline BMI [Mean (Standard Deviation); unit: Kg/m^2] | 22.38 (3.262) | 22.56 (3.497) | 22.52 (3.606) | 22.48 (3.448)
Baseline weight [Mean (Standard Deviation); unit: kg] | 63.5 (12.39) | 63.9 (12.88) | 64.0 (11.88) | 63.8 (12.34)
DSM-IV diagnosis of Schizophrenia [Count of Participants; unit: Participants]
  295.10 schizophrenia, disorganized type | 13 | 6 | 7 | 26
  295.30 schizophrenia, paranoid type | 88 | 81 | 85 | 254
  295.90 schizophrenia, undifferentiated type | 9 | 17 | 20 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6.
Description: PANNS total score: Changes from baseline over time - mixed model for repeated measures at week 6 -PANSS total score may range from 30 to 210- Higher values of PANSS total score represent greater severity of illness
  LS Mean and SE for change from baseline are based on Mixed Model for Repeated Measures with fixed effects terms for treatment, visit (as a categorical variable), pooled country, age strata, PANSS total score at baseline, and treatment-by-visit interaction.
Time Frame: Baseline to 6 weeks
Population: The ITT population includes all randomized subjects who receive at least one dose of study medication and have at least one post-baseline assessment in any efficacy variable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 94.5 (10.97) | 94.0 (11.12) | 92.8 (11.08)
  Week 6 | -18.6 (1.59) | -18.3 (1.60) | -10.5 (1.59)
Statistical Analysis 1: Comparison: Lurasidone 40 mg vs Placebo; The sample size was estimated to provide at least 85% power to reject at least one of the null hypotheses of no difference between placebo and lurasidone doses. LS Mean, LS mean difference, and the associated 95% CI and p-value for change from baseline are based on Mixed Model for Repeated Measures (MMRM); Test type: Superiority or Other; p = 0.0003, LS mean difference (SE); LS mean difference (SE) = -8.0, 95% CI 2-sided [-12.4 to -3.7]
Statistical Analysis 2: Comparison: Lurasidone 80 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0006, LS mean difference (SE); LS mean difference (SE) = -7.7, 95% CI 2-sided [-12.1 to -3.4]

2. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Scale
Description: Clinical Global Impression severity (CGI-S): Changes from baseline over time-mixed model for repeated measures- scale from 1-7 - 1=normal, not at all ill; 7=among the most extremely ill patients.
  LS Mean and SE for change from baseline are based on Mixed Model for Repeated Measures with fixed effects terms for treatment, visit (as a categorical variable), pooled country, age strata, CGIS at baseline, and treatment-by-visit interaction.
Time Frame: baseline, week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 4.9 (0.62) | 4.8 (0.66) | 4.8 (0.61)
  week 6 | -0.97 (0.093) | -0.92 (0.093) | -0.50 (0.094)
Statistical Analysis 1: Comparison: Lurasidone 40 mg vs Placebo; LS Mean, LS mean difference, and the associated 95% CI and p-value for change from baseline are based on Mixed Model for Repeated Measures (MMRM); Test type: Superiority or Other; p = 0.0003, LS mean difference (SE); LS mean difference (SE) = -0.47, 95% CI 2-sided [-0.73 to -0.22]
Statistical Analysis 2: Comparison: Lurasidone 80 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0015, LS mean difference (SE); LS mean difference (SE) = -0.42, 95% CI 2-sided [-0.67 to -0.16]

3. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Scores
Description: PANSS positive subscale score: changes from baseline over time - mixed model for repeated measures -Positive subscale (range 7-49): sum of Items P1 to P7 in the positive subscale - Higher values of PANSS Positive Subscale Score represent greater severity of illness
  LS Mean and SE for change from baseline are based on Mixed Model for Repeated Measures with fixed effects terms for treatment, visit (as a categorical variable), pooled country, age strata, corresponding PANSS subscale score at baseline, and treatment-by-visit interaction.
Time Frame: baseline, week 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 24.1 (3.96) | 24.0 (4.08) | 23.4 (3.75)
  week 6 | -6.3 (0.51) | -6.3 (0.51) | -3.1 (0.51)

4. Secondary Outcome: Change From Baseline in PANSS Positive, Negative Subscale Scores
Description: PANSS Negative subscale score: changes form baseline over time - Mixed model for repeated measures - - Negative subscale (range 7-49): sum of Items N1 to N7 in the negative subscale - Higher values of PANSS Negative Subscale Score represent greater severity of illness
  LS Mean and SE for change from baseline are based on Mixed Model for Repeated Measures with fixed effects terms for treatment, visit (as a categorical variable), pooled country, age strata, corresponding PANSS subscale score at baseline, and treatment-by-visit interaction.
Time Frame: baseline, week 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 24.2 (4.32) | 24.5 (4.37) | 24.4 (4.01)
  week 6 | -4.0 (0.48) | -3.8 (0.49) | -2.3 (0.49)

5. Secondary Outcome: Proportion of Responders, Where Response is Based on ≥ 20% Improvement From Baseline in PANSS Total Score at Week 6
Description: PANSS responder analysis over time: achieving >= 20% reduction from baseline
Time Frame: week 6
Population: ITT Population
Measure: Number; unit: number of participants
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
number of participants | 69 | 47 | 69

6. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q)
Description: PQ-LES-Q percentage maximum possible score: summary statistics over time - PQ-LES-Q % maximum possible score can range from 0% to 100%. Higher scores indicate better quality of life.
  LS Mean and SE for change from baseline are from an ANCOVA model including factors of treatment, pooled country and age group (stratification factor), and corresponding Baseline score as covariate and LOCF approach.
Time Frame: baseline, week 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 51.3 (17.26) | 53.6 (18.50) | 52.5 (15.67)
  week 6 | 5.6 (1.28) | 6.1 (1.30) | 0.3 (1.24)

7. Secondary Outcome: Change From Baseline in Clinician-rated Children's Global Assessment Scale (CGAS)
Description: Clinician-rated Children's Global Assessment Scale (CGAS) score: summary statistics over time - CGAS is a numeric scale (1 through 100) , where 1 represents the most impaired functioning and 100, superior functioning
  LS Mean and SE for change from baseline are from an ANCOVA model including factors of treatment, pooled country and age group (stratification factor), and corresponding Baseline score as covariate and LOCF approach.
Time Frame: baseline, week 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 44.2 (9.33) | 44.6 (8.11) | 43.9 (8.34)
  week 6 | 11.3 (1.16) | 11.9 (1.18) | 7.5 (1.17)

8. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Scores
Description: PANSS general psychopathology subscale score: changes from baseline over time - mixed model for repeated measures -- General psychopathology (range 16-112): sum of Items G1 to G16 in the general psychopathology subscale -Higher values of PANSS General Psychopathology Subscale Score represent greater severity of illness
  LS Mean and SE for change from baseline are based on Mixed Model for Repeated Measures with fixed effects terms for treatment, visit (as a categorical variable), pooled country, age strata, corresponding PANSS subscale score at baseline, and treatment-by-visit interaction.
Time Frame: baseline, week 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 46.2 (6.65) | 45.5 (7.03) | 45.0 (6.94)
  week 6 | -8.1 (0.80) | -8.1 (0.81) | -5.3 (0.80)

9. Secondary Outcome: Change From Baseline in PANSS Excitability Subscale Scores
Description: Excitability subscale scores (range 4-28): consists of the following four items from the PANSS: excitement, hostility, uncooperativeness, and poor impulse control
  * Higher values of PANSS Excitability Subscale Score represent greater severity of illness
  LS Mean and SE for change from baseline are based on Mixed Model for Repeated Measures with fixed effects terms for treatment, visit (as a categorical variable), pooled country, age strata, corresponding PANSS subscale score at baseline, and treatment-by-visit interaction.
Time Frame: baseline, week 6
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Number analyzed (Participants) | 108 | 106 | 112
units on a scale
  baseline | 10.8 (2.91) | 11.1 (3.07) | 10.7 (3.23)
  week 6 | -0.6 (0.33) | -1.7 (0.33) | -2.4 (0.33)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) is defined as an AE with a start date on or after the date of first dose through 7 days after study drug discontinuation (14 days for serious adverse events and deaths) for subjects who complete the double blind study but do not enter into the extension study or early discontinue during the double blind study), or through the last study day of the doubleblind period for subjects continuing into the extension study.
Description: AEs were collected from the time the informed consent is signed to the end of the study. Non-leading questions were used to ask subjects about the possible occurrence of AEs. The investigator then established a diagnosis of the event based on signed, symptoms, and/or other clinical information. Please note that two subjects from the lurasidone 80mg (originally 106) group transferred to the lurasidone 40 mg (originally 108) group
Arm/Group | Lurasidone 40 mg | Lurasidone 80 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/110 | 2/104 | 9/112
Other Adverse Events (participants affected / at risk) | 70/110 | 67/104 | 53/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 40 mg (N=110) | Lurasidone 80 mg (N=104) | Placebo (N=112)
schizophrenia (Psychiatric disorders) | 2 (2) | 2 (2) | 7 (7)
Homicidal Ideation (Psychiatric disorders) | 1 | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 40 mg (N=110) | Lurasidone 80 mg (N=104) | Placebo (N=112)
Somnolence (Nervous system disorders) | 10 (10) | 12 (12) | 6 (8)
Headache (Nervous system disorders) | 7 (8) | 11 (15) | 14 (19)
Akathisia (Nervous system disorders) | 10 (12) | 9 (10) | 2 (2)
Sedation (Nervous system disorders) | 6 (6) | 2 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 14 (20) | 15 (18) | 3 (4)
Vomiting (Gastrointestinal disorders) | 9 (10) | 7 (8) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6) | 7 (8) | 10 (12)
Agitation (Psychiatric disorders) | 5 (7) | 6 (6) | 5 (5)
Anxiety (Psychiatric disorders) | 11 (14) | 3 (3) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.